CLINICAL TRIAL: NCT03831373
Title: Effects of Resistance Exercise Focused on the Upper Body Versus the Lower Body on Global Physical Fitness and Cognitive Status of Older Adults Living in Geriatric Centers
Brief Title: Upper Versus Lower Body Resistance Exercise in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vigo (Other)
Responsible Party: Principal Investigator, Miguel A. Sánchez-Lastra, Principal Investigator, University of Vigo
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 16-1009-17
Record Dates: First submitted 2018-10-09; First posted 2019-02-05 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Quality of Life; Aging
Keywords: Exercise
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Upper-limb-focused resistance training (Experimental)
  Interventions: Other: Physical exercise
- Lower-limb-focused resistance training (Experimental): Lower-limb-focused resistance training with elastic bands.
  Interventions: Other: Physical exercise
- Stretching exercise (Active Comparator): Stretching exercise program in a sitting position.
  Interventions: Other: Physical exercise

INTERVENTIONS:
Other: Physical exercise — Three physical exercise programs, two of resistance training with elastic bands and one of stretching exercises, all performed in a sitting position.

SUMMARY:
TITLE: Relation between focused resistance training and its effect on cognitive performance and functional Independence of institutionalized elderly.

HIPOTHESIS: The performance of a physical exercise program based on resistance training in older adults stabilizes or improves some parameters of the functional independence as well as the cognitive function, finding effects overall organism by the focused training of some muscular groups.

GENERAL OBJECTIVES: 1) to analyze the differential effects of an exercise program based on the training of the muscular strength of the upper body versus a lower body one, at short and long term in institutionalized elderly people; 2) to identify if there is any relations between the variables that induce frailness or functional dependence and the physical exercise program.

SPECIFIC OBJECTIVES: To determine the differential effects of a physical exercise program based on the development of the muscular strength of the upper body versus the lower body, in sessions of 40 minutes a day, 2 days per week during 7 months on: a) The improvement of functional independence by the amelioration of balance, decrease of fall risk and an adequate development in the activities of daily living; b) The improvement of the global cognitive function; c) The improvement of the quality of life.

METHODS

* Design: Controlled trial. The institutionalized elderly from the geriatric centers will be invited to take part in the study. After they meet the selection criteria, they will be assigned to two experimental groups and one control group in each center. Information regarding sociodemographic characteristics and a clinical anamnesis of the participants will be collected.
* Intervention: Three groups, one from each centre. Two centers, experimental groups, will perform two physical exercises programs of resistance training with elastic bands, one focused on the upper and one on the lower body. They will be carried 2 days per week, during 3 months in 45-minute sessions. The program will consist of 5 exercises, with a volume of 4 sets of 12 repetitions, with 2-minute breaks between sets and 3 between exercises. Control group will participate in 40 minutes stretching sessions, 3 times per week. After 3 months of exercise and after three months of transition, they experimental groups will perform the other program for another 3 months, crossing the interventions.
* Assessments: Six will be carried: At the beginning, at the end of the first intervention, at the beginning of the second one, at the end and a follow up 3 months later. In each, it will be assessed the potential cognitive impairment and cognitive status (Spanish version of the MMSE, Fototest and Trail Making Test part A), functional independence (Timed Up and Go Test), grip strength (hand dynamometer), lower body strength (30 Seconds Chair Stands) and flexibility/mobility (Chair Sit-and-Reach and Back Scratch Test.)

ELIGIBILITY:
Inclusion Criteria:

* No medical contraindications to be involved in the exercise programs.
* To be able to follow the exercise classes
* Signed informed consent

Exclusion Criteria:

-

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2018-02-21 (Actual); Primary Completion 2019-03-21 (Actual); Study Completion 2019-03-21 (Actual)

PRIMARY OUTCOMES:
Spanish version of the Mini-Mental State Examination. | 24 weeks
  The Mini-Mental State Examination is a 30-point questionnaire comprised by eight different categories and score range. Orientation to time (0-5 points) Orientation to place (0-5 points) Registration (0-3 points) Attention and calculation (0-5 points) Recall (0-3 points) Language (0-2 points) Repetition (0-1 points) Complex commands (0-6 points). Interpretation: Any score greater than or equal to 24 points (out of 30) indicates a normal cognition. ≤9 points: severe cognitive impairment 10-18 points: moderate cognitive impairment and 19-23 points: mild cognitive impairment.
Test of the pictures | 24 weeks
  The test of the pictures (Fototest in the Spanish version) is used to assess the short and long-term memory, the verbal fluency and denomination capacities. The test is well correlated with the Mini-mental State Examination and it's reference values are situated in 34.4±4.4.
Trail Making Test part A. | 24 weeks
  The Trail Making Test part A. The time required by an individual to draw lines sequentially connecting 25 encircled numbers distributed on a sheet of paper is measured.
Timed Up and Go Test | 24 weeks
  Standardized test to assess the basic functional mobility of elderly persons. The patient is observed and timed while he rises from an arm chair, walks 3 meters, turns, walks back, and sits down again.
Grip Strength | 24 weeks
  Assessed by means of a hand-held dynamometer, Grip Strength: By means of a hand-held dynamometer, this assessment has been stated as a predictor of frailty and mortality.
Chair Sit and Reach | 24 weeks
  Present in the Senior Fitness Test, to assess the mobility/flexibility of the lower back and limbs.
Back Scratch Test | 24 weeks
  Present in the Senior Fitness Test, this evaluates the joint mobility of the shoulders.

CONTACTS AND LOCATIONS:
Locations (1):
- DomusVi Barreiro, Vigo, Galicia, Spain

REFERENCES:
- [Derived] Sanchez-Lastra MA, Varela S, Cancela JM, Ayan C. Upper versus lower body resistance exercise with elastic bands: effects on cognitive and physical function of institutionalized older adults. Eur Geriatr Med. 2022 Aug;13(4):907-916. doi: 10.1007/s41999-022-00616-6. Epub 2022 Feb 12. PMID 35150433